CLINICAL TRIAL: NCT06954883
Title: Effectiveness of Augmented Reality as a Distraction Technique for Reducing Pain and Anxiety in Pediatric Dental Extractions: A Parallel-Group, Double-Blind Randomized Controlled Trial
Brief Title: Augmented Reality Distraction for Reducing Pain in Pediatric Dental Procedures
Acronym: AR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ِAhmed kamel Abdel Naser soliman, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-2024-0004
Record Dates: First submitted 2025-04-08; First posted 2025-05-02 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized controlled trial with a 1:1 allocation ratio. Participants were randomized into either the experimental group (augmented reality distraction during dental procedures) or the control group (standard tell-show-do technique). Each participant received only one of the two interventions. No crossover occurred between groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessors/data analysts don't know group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR Distraction (Experimental): Participants wear AR/VR goggles showing an interactive cartoon during LA injection and extraction.
  Interventions: Behavioral: Augmented Reality Distraction
- Tell-Show-Do (Active Comparator): Participants undergo standard Tell-Show-Do behavior guidance during treatment.
  Interventions: Behavioral: Standard Care (Tell-Show-Do Technique)

INTERVENTIONS:
Behavioral: Augmented Reality Distraction — Participants in this group wore augmented reality (AR) goggles during local anesthesia administration and dental extraction. The AR system displayed interactive 3D animated videos (celestial bodies) to divert attention and reduce procedural pain and anxiety.
  Arms: AR Distraction
Behavioral: Standard Care (Tell-Show-Do Technique) — Children aged 6-10 years (both sexes, Egyptian ethnicity) received behavioral management using the Tell-Show-Do (TSD) technique during primary anterior tooth extraction under local infiltration anesthesia. The clinician explained the procedure in child-friendly language (Tell), demonstrated instruments in a non-threatening manner (Show), and then performed the extraction (Do) without augmented reality or audiovisual distraction.
  Arms: Tell-Show-Do

SUMMARY:
This randomized controlled trial evaluates the effectiveness of augmented reality (AR) as a distraction technique to reduce procedural pain and anxiety in children aged 6-10 undergoing primary tooth extraction. Participants will be randomly assigned to receive either AR distraction via VR goggles or standard tell-show-do behavior management during local anesthesia administration and extraction.

DETAILED DESCRIPTION:
Pain and anxiety are major challenges in pediatric dental care. AR presents an innovative, non-pharmacological technique to manage procedural distress. The study compares AR distraction versus conventional behavioral guidance in terms of self-reported pain (Wong-Baker FACES), dental anxiety (CFSS-DS), and physiological anxiety (heart rate monitoring). A double-blind design will ensure unbiased outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-10 years

Indicated for anterior primary tooth extraction

No previous exposure to local anesthesia

Exclusion Criteria:

* Medically compromised children

Children with cognitive or communication impairments

Children who underwent similar treatment within the past 3 months

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Status: Completed Actual Enrollment: 60 participants Start Date: May 15 2025 Primary Completion Date: July 30 2025 Study Completion Date: August 15 2025
  Recruitment Locations:
  • Faculty of Dentistry, Assuit University, Egypt
  Eligibility Criteria:
  * Ages: 6-10 years
  * Sex: All
  * Accepts Healthy Volunteers: Yes
  * Inclusion Criteria:
    * Children requiring primary anterior tooth extractions
    * No prior experience of local anesthesia
  * Exclusion Criteria:
    * Previous local anesthesia
Pre-assignment Details: Number of Participants Screened: 60 eligible participants were enrolled after screening
  Reasons for Exclusions:
  * previous anesthesia experience, special needs, anxiety disorder diagnosis, recent root planing)
  * Declined to participate
  Number Assigned to Arms:
  * AR Group: 30 participants
  * Control Group: 30 participants
Groups:
- AR-based Distraction: Children aged 6-10 years (both sexes, Egyptian ethnicity) received augmented reality (AR) distraction during primary anterior tooth extraction under local infiltration anesthesia. Each child selected a cartoon video displayed through a head-mounted AR/VR device (IGY 360 headset connected to a smartphone). The device projected AR animations (e.g., 3D celestial bodies) into the child's view, diverting attention throughout topical anesthesia, injection, and extraction.
Period: Overall Study
Arm/Group | AR-based Distraction | Standard Care (Tell-Show-Do Technique)
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (N=60; AR group n=30, Control group n=30) were included in baseline analyses. No participants were excluded after randomization, and baseline data were complete for all individuals.
Groups:
- AR-based Distraction: Children aged 6-10 years (both sexes, Egyptian ethnicity) received augmented reality (AR) distraction during primary anterior tooth extraction under local infiltration anesthesia. Each child selected a cartoon video displayed through a head-mounted AR/VR device (IGY 360 headset connected to a smartphone). The device projected AR animations (e.g., 3D celestial bodies) into the child's view, diverting attention throughout topical anesthesia andinjection.
- Total: Total of all reporting groups
Arm/Group | Standard Care (Tell-Show-Do Technique) | AR-based Distraction | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years at the time of enrollment, measured as the difference between the participant's date of birth and the date of study enrollment. Reported as mean ± standard deviation (SD) in years Units: Years (mean and SD)
  Years | 7.9 (1.1) | 7.8 (1.2) | 7.85 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Biological sex of participants as reported by the parent or legal guardian at enrollment. Categorized as male or female and reported as number and percentage of participants in each arm.
  Units: Number (%)
  Participants
    Female | 15 | 14 | 29
    Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
CFSS-DS [Mean (Standard Deviation); unit: score on a scale] — Dental anxiety was assessed before the procedure using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS). The CFSS-DS is a validated 15-item questionnaire scored on a 5-point Likert scale (1 = not afraid to 5 = very afraid; total range 15-75, higher scores = greater anxiety). Values were compared between study arms (Augmented Reality distraction vs. Standard Care)
  score on a scale | 30.1 (5.2) | 29.7 (4.8) | 29.9 (4.97)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Heart rate was measured in beats per minute (bpm) using a finger pulse oximeter (CMS 50DL, China). Measurements were taken while the child was seated in the dental chair before the procedure as a physiological indicator of anxiety. Values are reported as mean ± standard deviation (SD). The outcome was defined as the post-procedure heart rate value, compared between study arms.
  beats per minute | 94 (11) | 95 (10) | 94.5 (10.43)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Using Wong-Baker FACES Scale
Description: Pain was assessed immediately after local anesthesia injection using the Wong-Baker FACES Pain Rating Scale. This validated pediatric pain scale consists of six facial expressions ranging from 0 ("No pain") to 10 ("Worst pain"). Children were asked to select the face that best represented their pain experience, which was then converted into a numeric score. Values are reported as mean ± standard deviation (SD)and were compared between study arms.
Time Frame: Immediately after the dental extraction procedure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AR-based Distraction | Standard Care (Tell-Show-Do Technique)
Number analyzed (Participants) | 30 | 30
Score on a scale | 2.3 (1.2) | 4.5 (1.3)

2. Secondary Outcome: 1. Children's Fear Survey Schedule-Dental Subscale
Description: Dental anxiety was assessed immediately post-procedure using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS). The CFSS-DS is a validated 15-item questionnaire scored on a 5-point Likert scale (1 = not afraid to 5 = very afraid; total range 15-75, higher scores = greater anxiety). Values were compared between study arms (Augmented Reality distraction vs. Standard Care)
Time Frame: Immediately after the dental extraction procedure.
Population: The analysis population consisted of all enrolled and randomized children who completed the CFSS-DS questionnaire immediately after the dental extraction procedure (N = 60; AR-based Distraction n = 30, Standard Care n = 30). No exclusions occurred and complete data were available for all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR-based Distraction | Standard Care (Tell-Show-Do Technique)
Number analyzed (Participants) | 30 | 30
score on a scale | 17.6 (3.9) | 26.8 (4.5)

3. Secondary Outcome: Heart Rate as Physiological Indicator of Anxiety
Description: Heart rate was measured in beats per minute (bpm) using a finger pulse oximeter (CMS 50DL, China). Measurements were taken while the child was seated in the dental chair immediately post-procedure as a physiological indicator of anxiety. Values are reported as mean ± standard deviation (SD). The outcome was defined as the post-procedure heart rate value, compared between study arms.
Time Frame: Immediately post-procedure
Population: All randomized participants were included in the analysis of heart rate (N = 60; AR-based Distraction n = 30, Standard Care n = 30). No participants were excluded and no data were missing.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | AR-based Distraction | Standard Care (Tell-Show-Do Technique)
Number analyzed (Participants) | 30 | 30
beats per minute (bpm) | 80 (8) | 89 (10)

ADVERSE EVENTS:
Time Frame: From the start of the dental extraction procedure until 1 hour post-procedure."
Description: Adverse events were defined broadly as any undesirable experience reported by the child or observed by the dental team during or after the extraction procedure. The focus was on minor, short-term reactions potentially related to the AR headset (e.g., dizziness, headache, eye strain) or the dental extraction (e.g., mild bleeding, transient discomfort). Events were recorded only if they occurred during the dental visit or within 1 hour post-procedure.
Arm/Group | AR Distraction | Tell-Show-Do
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This study was limited by its relatively small sample size and single-center setting, which may affect generalizability. Outcomes were assessed only immediately after the procedure, without longer-term follow-up."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT06954883/Prot_SAP_000.pdf